CLINICAL TRIAL: NCT03457831
Title: Status Epilepticus in the Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Ictal Group (Other)
Collaborators: Versailles Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICTAL SE REGISTRY
Record Dates: First submitted 2018-02-28; First posted 2018-03-08 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Status Epilepticus: Convulsive and Non-Convulsive Status Epilepticus ; and Pseudo Status Epilepticus

SUMMARY:
Convulsive and Non Convulsive Status Epilepticus (SE) and Pseudo Status Epilepticus prospective registry.

Data collection using a standardized form : demographic data and data related to the SE, including circumstances of onset, dates and times of onset and of seizure control, on-scene clinical findings, clinical features of the seizures, pre-hospital and hospital care providers, timing of antiepileptic and supportive treatments, results of etiological investigations, cause of SE, type and dosage of antiepileptic drugs. Dates and times of EEG monitoring, EEG results. Outcomes including vital status and Glasgow Outcome Scale score at ICU and hospital discharge, day-90 and 1-year after SE and determined based on data in the ICU and/or neurologist charts and/or patients phone interview.

ELIGIBILITY:
Inclusion Criteria:

* SE defined as 5 min or more of (i) continuous clinical and/or electrographic seizure activity or (ii) recurrent seizure activity without recovery (returning to baseline) between seizures.
* age >= 18 years

Exclusion Criteria:

* age < 18 years
* postanoxic status epilepticus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: critically ill patients requiring ICU hospitalisation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome | 1 year
  A favorable outcome is defined by a Glasgow Outcome Scale (GOS) of 5. The Glasgow Outcome Scale (GOS) will be determined according to patients charts review and/or general practitioner interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]

SECONDARY OUTCOMES:
Favorable outcome | 3 months, 5-years and 10 years
  A favorable outcome is defined by a Glasgow Outcome Scale (GOS) of 5. The Glasgow Outcome Scale (GOS) will be determined patients charts review and/or general practitioner interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]
Functional impairment | 3 months, and 1-year, 5-years and 10-years
  Percentages of the patients that experience functional impairment (motor, sensitive, cognitive, epilepsy)
total seizure duration | 72 hours
  total seizure duration in minutes
percentages of the patients that experience recurrent convulsive and/or non-convulsive seizures within 12 hours after ICU admission | 12 hours
refractory status epilepticus | 24 hours
super refractory status epilepticus | 72 hours
total ICU and in-hospital length of stay | 90 days
  total ICU and in-hospital length of stay in days
mortality rate | ICU and hospital discharge, 3-months, and 1-year, 5 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: stephane LEGRIEL, MD, Principal Investigator — Ictal Group
Locations (20):
- France (20):
  - CH Angouleme - Service de réanimation polyvalente, Angoulême
  - CH de Beauvais - Service de réanimation polyvalente, Beauvais
  - CH de Bethune - Service de Réanimation et Surveillance continue, Beuvry
  - Centre Hospitalier Universitaire Régional, Brest
  - CH Brive La Gaillarde - Service de réanimation - USC, Brive-la-Gaillarde
  - CH de Cannes, Cannes
  - CH Public du Cotentin - Service de Réanimation - Médecin intensive, Cherbourg
  - CHU Beaujon, Clichy
  - Hopitaux Universitaires Henri Mondor - Service d'anesthésie et des réanimations chirurgicales, Unité d'anesthésie-réanimation chirurgical cardiovasculaire, Créteil
  - Centre Hospitalier de Dieppe, Dieppe
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - CH de La Rochelle - Service de réanimation - USC, La Rochelle
  - Intensive Care Unit - Versailles Hospital, Le Chesnay
  - Hôpital privé Jacques Cartier - Service de réanimation médico chirurgicale, Massy
  - Groupe Hospitalier Sud Ile de France - Service de Réanimation - Médecin intensive, Melun
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Groupe Hospitalier Paris Saint Joseph - Service de réanimation médico chirurgicale, Paris
  - HP Claude Galien - Service de Réanimation Polyvalente, Quincy-sous-Sénart
  - Centre hospitalier de Roanne - Service de Réanimation - Soins continus, Roanne
  - Centre Hospitalier de Toulon, Toulon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vieille T, Jacq G, Merceron S, Huriaux L, Chelly J, Quenot JP, Legriel S. Management and outcomes of critically ill adult patients with convulsive status epilepticus and preadmission functional impairments. Epilepsy Behav. 2023 Apr;141:109083. doi: 10.1016/j.yebeh.2023.109083. Epub 2023 Feb 18. PMID 36803873
- [Derived] Chinardet P, Gilles F, Cochet H, Chelly J, Quenot JP, Jacq G, Soulier P, Lesieur O, Beuret P, Holleville M, Bruel C, Bailly P, Sauneuf B, Sejourne C, Galbois A, Fontaine C, Perier F, Pichon N, Arrayago M, Mongardon N, Schnell D, Lascarrou JB, Convers R, Legriel S. Electrocardiographic Changes at the Early Stage of Status Epilepticus: First Insights From the ICTAL Registry. Crit Care Med. 2023 Mar 1;51(3):388-400. doi: 10.1097/CCM.0000000000005768. Epub 2022 Dec 19. PMID 36533915
- [Derived] Jacq G, Chelly J, Quenot JP, Soulier P, Lesieur O, Beuret P, Holleville M, Bruel C, Bailly P, Sauneuf B, Sejourne C, Rigaud JP, Galbois A, Arrayago M, Plantefeve G, Stoclin A, Schnell D, Fontaine C, Perier F, Bougouin W, Pichon N, Mongardon N, Ledoux D, Lascarrou JB, Legriel S. Multicentre observational status-epilepticus registry: protocol for ICTAL. BMJ Open. 2022 Feb 15;12(2):e059675. doi: 10.1136/bmjopen-2021-059675. PMID 35168989